CLINICAL TRIAL: NCT05842525
Title: The Efficacy and Safety of Fruquintinib Plus FOLFIRI as Second-line Treatment in RAS-mutated Metastatic Colorectal Cancer
Brief Title: Fruquintinib Plus FOLFIRI in RAS-mutated Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hunan Cancer Hospital (Other)
Collaborators: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNSZL-FK-01
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer
Keywords: Fruquintinib; RAS-mutant; second-line
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Opiate Substitution Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): Fruquintinib combined with FOLFIRI
  Interventions: Drug: intensive treatment; Drug: Maintenance treatment

INTERVENTIONS:
Drug: intensive treatment — Fruquintinib 4mg, orally, once daily, 3 weeks on/ 1 week off Irinotecan 150 mg/m2 LV 400 mg/m2 5-fluorouracil 400mg/m2 and a 46-48h continuous infusion 2400mg/m2 on day 1, q2w （intensive treatment up to 8 cycels）
Drug: Maintenance treatment — Fruquintinib 5mg, orally, once daily, 3 weeks on/ 1 week off

SUMMARY:
RAS mutations are found in nearly half of colorectal cancer patients. However, except for G12C mutation, no driven gene targeted drug can be used. the commonly first-line used treatment regimen is bevacizumab combined with chemotherapy. Angiogenesis is an important therapeutic target in colorectal carcinoma. Fruquintinib is an oral small molecule inhibitor of VEGFR1/2/3, has approved for the third-line treatment of refractory colorectal cancer.

DETAILED DESCRIPTION:
This is a prospective ,single-center, open labeled, single-arm phase II study exploring the efficacy and safety of fruquintinib combined with FOLFIRI as second-line treatment of RAS-mutated metastatic colorectal cancer (mCRC) in patients with disease progression during or after first-line therapy with bevacizumab, oxaliplatin, and a fluoropyrimidine.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmed colorectal cancer;
2. RAS mutation;
3. Expected survival >12 weeks;
4. Patients had disease progression during or within 3 months of the last dose of first-line therapy, which must include bevacizumab combined with oxaliplatin, and a fluoropyrimidine;
5. ECOG PS 0-1;
6. At least one measurable lesion (according to RECIST1.1);
7. Adequate hepatic, renal, heart, and hematologic functions;
8. Negative serum pregnancy test at screening for women of childbearing potential.

   -

Exclusion Criteria:

1. MSI-H / dMMR;
2. Received radiation therapy, surgical procedure, immunotherapy or other investigational drugs within 4 weeks prior to treatment ;
3. Prior treatment with anti-angiogenic small molecule targeted drugs, such as fruquintinib, etc;
4. Prior treatment with an irinotecan-based chemotherapy regimen;
5. Symptomatic brain or meningeal metastases (except for patients with BMS who have received local radiotherapy or surgery for more than 6 months and whose disease is stable);
6. Severe infection (e.g., requiring intravenous antibiotics, antifungal drugs, or antiviral drugs) within 4 weeks prior to treatment;
7. Patients with hypertension that cannot be well controlled by antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
8. Patients who had active bleeding or coagulopathy within 2 months before enrollment, had a tendency to bleed, or were receiving thrombolytic therapy and were considered by the investigator to be ineligible for enrollment;
9. Active heart disease, including myocardial infarction, severe/unstable angina, 6 months prior to treatment. Echocardiography examination left ventricular ejection fraction < 50%, arrhythmia control is not good;
10. The patient has had other malignant tumors within 5 years (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix); Allergy to the study drug or any of its excipients;
11. The patient is unable to take the drug orally, or the patient has a condition judged by the investigator to affect the absorption of the drug; Women who are pregnant (with a positive pregnancy test before medication) or breastfeeding;
12. Urine routine showed urine protein ≥2+, and 24-hour urine protein level >1.0g; Other conditions deemed by the investigator to be ineligible for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-05-28 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | assessed up to 1 year
  the proportion of patients with complete response or partial response, using RECIST v 1.1

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | assessed up to 1 year
  time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first.
  Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator

OTHER OUTCOMES:
Overall survival (OS) | assessed up to 2 year
  time from randomization to death from any cause.
Disease Control Rate (DCR) | assessed up to 1 year
  the proportion of patients with complete response, partial response or stable disease, using RECIST v 1.1

CONTACTS AND LOCATIONS:
Overall Officials: zhenyang Liu, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No